CLINICAL TRIAL: NCT05073029
Title: Personalized Nutrition, Physical Activity and Therapy to Modulate Gut Microbiota: a Randomized Clinical Study to Promote a Healthy Lifestyle in Students
Brief Title: Open Label Randomized Clinical Study to Promote a Healthy Lifestyle in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Collaborators: Taras Shevchenko National University of Kyiv (Other)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor, Endocrinology Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ENDO-7
Record Dates: First submitted 2021-10-08; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Healthy; Obesity; Nutrition, Healthy; Vitamin D Deficiency
Keywords: gut microbiota; vitamin D; personalized nutrition; lifestyle in students; synbiotic; depression
MeSH Terms: conditions — Obesity; Vitamin D Deficiency; Depression | interventions — Synbiotics; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care group (Active Comparator): 3-month course of individually selected nutrition program developed by a gastroenterologist-nutritionist and modification of physical activity (8000-10000 steps daily)
  Interventions: Other: nutrition program and modification of physical activity
- intervention group (Experimental): additionally to previous group recieved treatment with synbiotic (Fructooligosaccharides+Lactobacillus rhamnosus GG ATCC 53103) and vitamin D3 - 2000 IU. The students were instructed to take vitamin D3 and synbiotic sachets twice a day for 3 months.
  Interventions: Dietary Supplement: synbiotic (Fructooligosaccharides+Lactobacillus rhamnosus GG ATCC 53103, 4.0х109 colony forming units - CFU); Dietary Supplement: vitamin D3

INTERVENTIONS:
Other: nutrition program and modification of physical activity — nutrition program developed by a gastroenterologist-nutritionist and modification of physical activity (8000-10000 steps daily)
  Arms: standard care group
Dietary Supplement: synbiotic (Fructooligosaccharides+Lactobacillus rhamnosus GG ATCC 53103, 4.0х109 colony forming units - CFU) — one synbiotic sachet (3g), BID, for 3 month traetment
  Other Names: Acidolac
  Arms: intervention group
Dietary Supplement: vitamin D3 — vitamin D3, oral, 2000IU BID, for 3 month treatment
  Other Names: Olidetrim
  Arms: intervention group

SUMMARY:
The main medical and social purpose of the project "It's trendy to be healthy!" is the promotion of healthy lifestyles and healthy eating among student youth. The relevance of this project is beyond doubt, as the WHO called obesity a non-communicable epidemic, and according to research by the Jane Schiller University of Germany (Germany), as mentioned above, Ukraine topped the list of the countries with high mortality due to malnutrition

ELIGIBILITY:
Inclusion Criteria:

* medical students aged between 18-25 years;
* presence of presence of vitamin D deficiency or insuficiency (serum total vit D3 level less than );
* signed informed consent.

Exclusion Criteria:

* regular intake of probiotics, prebiotics, antibiotics, anticonvulsants, calcium and vit. D supplements for 3 months prior the inclusion;
* previously diagnosed allergy to gut microbiota-based therapy; gastrointestinal disorders including food allergy, gluten-sensitive enteropathy, ulcerative colitis;
* suffering from any psychiatric illness; presence of diabetes mellitus, chronic cardiovascular or respiratory disease, an active malignant tumor or chronic infections; participation in another clinical trial;
* pregnancy or lactation;
* any condition thought to be associated with poor compliance (e.g., alcoholism or drug addiction) or any condition or circumstance that would, in the opinion of the investigator, prevent completion of the study or interfere with analysis of study results.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Changes in Rathus Assertiveness Schedule | 90 days compared to baseline
  RAS is consists of 30 questions and is divided into five subgroups, according to the scores: 0-24: very insecure; 25-48: rather unsure than confident; 49-72: average confidence value; 73-96: self-confident and 97-120: overconfident.
Changes in test "Diagnosis of situational and personal anxiety" | 90 days compared to baseline
  Test " Diagnosis of situational and personal anxiety" by Ch. D. Spielberger consists of 20 statements that refer to anxiety as a state (state of anxiety, reactive (RA) or situational anxiety (SA)) and 20 statements to define anxiety as a disposition, personality traits (anxiety property).

SECONDARY OUTCOMES:
weight | at 45 and 90 days compared to baseline
  weight in kg
waist circumferences (WC) | at 45 and 90 days compared to baseline
  WC in cm
body mass index (BMI) | at 45 and 90 days compared to baseline
  weight in kg and height in meters will be combined to report BMI in kg/m^2
muscle mass | at 45 and 90 days compared to baseline
  muscle mass (kg) using electronic scales-analyzers of body composition Tanita Scale BC-601
fat content | at 45 and 90 days compared to baseline
  fat content (%) using electronic scales-analyzers of body composition Tanita Scale BC-601
systolic blood pressure (SBP) | at 45 and 90 days compared to baseline
  Blood pressure is measured from the right hand while sitting with the help of a mercury barometer "OMRON". Blood pressure is taken twice at a 5-minute interval while seated for 5 minutes.
diastolic blood pressure (DBP) | at 45 and 90 days compared to baseline
  Blood pressure is measured from the right hand while sitting with the help of a mercury barometer "OMRON". Blood pressure is taken twice at a 5-minute interval while seated for 5 minutes.
HbA1c | 90 days compared to baseline
  HbA1c in %
fasting plasma glucose (FPG) | 90 days compared to baseline
  FPG in mmol/L
total cholesterol (TC) | 90 days compared to baseline
  TC in mmol/L
Total vitamin D3 | 90 days compared to baseline
  Total vitamin D3, ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Nataliia Molochek, PhD, Study Director — ESC "Institute of Biology and Medicine", Taras Shevchenko National University of Kyiv; Liudmyla Ostapchenko, Professor, Study Chair — ESC "Institute of Biology and Medicine", Taras Shevchenko National University of Kyiv
Locations (2):
- Ukraine (2):
  - Bogomolets National Medical University, Kyiv
  - Taras Shevchenko National University of Kyiv, Kyiv

IPD SHARING:
Plan to Share IPD: No